CLINICAL TRIAL: NCT01429792
Title: A Multi-Center Study Evaluating the Rate of Genotype 1, 2, 3 & 4 Chronic Hepatitis C Patients With Slow Response / Non-rapid Viral Response to Anti-Viral Treatment of Pegasys (Peginterferon Alfa 2a) in Combination With Copegus (Ribavirin)
Brief Title: A Study Evaluating Slow Response/Non-Rapid Response in Patients With Chronic Hepatitis C, Genotype 1, 2, 3 & 4 Treated With Pegasys (Peginterferon Alfa-2a) and Copegus (Ribavirin)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21779
Record Dates: First submitted 2011-09-05; First posted 2011-09-07 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2017-12

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — standard treatment, subcutaneously weekly
Drug: ribavirin [Copegus] — standard treatment, orally daily

SUMMARY:
This multi-center study will evaluate the viral response in patients with chronic hepatitis C, genotype 1, 2, 3 & 4 on standard anti-viral treatment with Pegasys (peginterferon alfa-2a) and Copegus (ribavirin). Patients will receive weekly subcutaneous Pegasys plus daily oral Copegus for 24 weeks (genotype 2 & 3) or 48 weeks (genotype 1 & 4). Patients identified as slow responders/non-rapid virological responders will be eligible for an additional 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Serologic evidence of chronic hepatitis C, genotype 1, 2, 3 or 4 by anti-HCV antibody test
* Documented pre-treatment HCV RNA quantitative result
* Compensated liver disease (Child-Pugh Grade A)
* Patient receiving standard combination treatment of Pegasys (peginterferon alfa-2a and Copegus (ribavirin)

Exclusion Criteria:

* Decompensated liver disease (Child-Pugh Class B or C cirrhosis)
* Co-infection with active hepatitis A and/or hepatitis B
* History or evidence of a medical condition associated with liver disease other than HCV
* Signs and symptoms of hepatocellular carcinoma
* History of poorly controlled thyroid disease, elevated TSH or any clinical manifestations of thyroid disease
* Therapy with antineoplastic treatment </= 6 months prior to study day
* Diabetes mellitus in subjects receiving an insulin therapy
* Evidence of severe retinopathy
* Pregnant or breast-feeding women, and male partners of women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2008-09-25 (Actual); Primary Completion 2013-06-10 (Actual); Study Completion 2013-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- Israel (26):
  - Haemek Hospital; Gastroenterology, Afula
  - Clalit City Ashdod MC; Liver Clinic, Ashdod
  - Barzilai MC; Gastroenterology, Ashkelon
  - Batyamon; Liver Unit, Bat Yam
  - Soroka Medical Center; Liver Unit, Beersheba
  - Soroka Medical Center; Gastroenterology, Beersheba
  - Rambam Medical Center; Gastroenterology - Liver Unit, Haifa
  - Bnei-Zion Medical Center; Gastroenterology, Haifa
  - Carmel Hospital; Liver Unit, Haifa
  - Wolfson Hospital; Gastroenterology Unit, Holon
  - Hadassah Hospital; Liver Unit, Jerusalem
  - Clalit Strauss MC, Jerusalem
  - Meir Medical Center; Gastroenterology, Kfar Saba
  - Naharyia / Western Galilee MC; Gastro Unit, Nahariya
  - Holy Family Medical Center; Gastroenterology, Nazareth
  - Rabin Medical Center; Gastroenterology - Liver Unit, Petah Tikva
  - Hasharon Mc; Gastroenterology, Petah Tikva
  - Chaim Sheba Medical Center; Gastroenterology, Ramat Gan
  - Kaplan Medical Center; Gastroenterology Unit, Rehovot
  - Clalit Pinsker Rishon; Liver Clinic, Rishon LeZiyyon
  - Rebecca Sieff; Gastroenterology, Safed
  - Sourasky / Ichilov Hospital; Gastroenterology - Liver Unit, Tel Aviv
  - Clalit Zamenhoff, Tel Aviv
  - Maccabi Health Services MC, Tel Aviv
  - Poria Hospital; Gastroenterology, Tiberias
  - Assaf Harofeh; Gastroenterology, Ẕerifin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants, 18 years of age and above with serologically proven genotype 1, 2, 3 or 4 CHC and treated with the standard combination treatment of peginterferon alfa-2a (Pegasys) and ribavirin (Copegus).
Pre-assignment Details: A total of 1013 participants were enrolled in the study and 607 of them completed the study.
Groups:
- Pegylated Interferon Alfa 2a (Peginterferon): Participants with chronic hepatitis C (CHC) were treated with subcutaneous pegylated interferon once weekly in combination with ribavirin once daily.
Period: Overall Study
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Started | 1013
Genotype 1 | 687
Genotype 2 & 3 | 305
Genotype 4 | 5
Completed | 607
Not Completed | 406
Not completed — Other Reasons | 67
Not completed — Unknown Disposition | 94
Not completed — Negative HCV-RNA at Week 4 | 1
Not completed — Negative HCV-RNA at Week 12 | 4
Not completed — Decrease of less than 2-log in HCV RNA | 32
Not completed — Positive HCV-RNA at Week 24 | 50
Not completed — Withdrawal by Subject | 70
Not completed — Lost to Follow-up | 88

BASELINE CHARACTERISTICS:
Population: All participants who enrolled in the study
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Number analyzed (Participants) | 1013
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (11.3)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 380
  Male | 632
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Partial Early Virological Response (pEVR) to Study Treatment
Description: The rate of participants with pEVR to study treatment was defined as ≥ 2 log reduction in HCV-RNA level from baseline value to Week 12 of study treatment but with detectable HCV-RNA at Week 12.
Time Frame: Week 12
Population: Participants with CHC Genotype 1 & 4 at week 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Number analyzed (Participants) | 692
Percentage of participants | 15.7 [12.6 to 18.1]

2. Primary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR) to Study Treatment
Description: The rate of participants with a cEVR to study treatment was defined as negative HCV-RNA level at Week 12 of study treatment
Time Frame: Week 12
Population: Participants with CHC Genotype 1 & 4 at Week 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Number analyzed (Participants) | 692
Percentage of participants | 50.8 [46.8 to 54.4]

3. Primary Outcome: Percentage of Participants With Undetectable HCV-RNA at End of Treatment Response (ETR) at Week 24
Description: The rate of participants with undetectable HCV-RNA at ETR at Week 24 was defined as at least a 2-log decrement in HCV-RNA from the start of treatment, but with detectable HCV-RNA at Week 12 of study treatment and undetectable HCV-RNA at Week 24 of study treatment
Time Frame: Week 24
Population: Participants with CHC Genotype 1 & 4 at Week 24
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Number analyzed (Participants) | 456
Percentage of participants | 15.6 [12.9 to 19.2]

4. Primary Outcome: Percentage of Participants With Rapid Virologic Response (RVR) at Week 4
Description: The rate of participants with RVR was defined as negative HCV-RNA level at Week 4 of study treatment.
Time Frame: Week 4
Population: Participants with CHC Genotype 2 & 3 at Week 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Number analyzed (Participants) | 304
Percentage of participants | 48.03 [42.3 to 53.6]

5. Primary Outcome: Percentage of Participants Without a RVR (Non-RVR) at Week 4 of Standard Treatment
Description: The rate of participants without a RVR (non-RVR) was defined as detectible HCV-RNA level at Week 4 of standard treatment.
Time Frame: Week 4
Population: Participants with CHC Genotype 2 & 3 at Week 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Number analyzed (Participants) | 304
Percentage of participants | 51.97 [46.2 to 57.6]

6. Primary Outcome: Percentage of Participants With Non-RVR and Undetectable HCV-RNA at Week 24
Description: The rate of participants with non-RVR and undetectable HCV-RNA at Week 24 was defined as detectable HCV-RNA level at Week 4 of study treatment and undetectable HCV-RNA at Week 24 of study.
Time Frame: Week 24
Population: Participants with CHC Genotype 2 & 3 at Week 24
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Number analyzed (Participants) | 305
Percentage of participants | 6.9 [4.3 to 10.3]

7. Secondary Outcome: Percentage of Participants With pEVR to Study Treatment at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: As pre-specified in the protocol, genotypes 1 and 4 were combined due to insufficient enrollment for genotype 4.
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Number analyzed (Participants) | 0

8. Secondary Outcome: Percentge of Participants With a cEVR to Study Treatmen at Week 12 of Study Treatment
Description: as for outcome 2
Time Frame: Week 12
Population: As pre-specified in the protocol, genotypes 1 and 4 were combined due to insufficient enrollment for genotype 4.
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Participants With Undetectable HCV-RNA at Week 24, But With Detectable HCV-RNA atWeek 12 and Undetectable HCV-RNA at Week 24
Description: as for outcome 3
Time Frame: Week 24
Population: As pre-specified in the protocol, genotypes 1 and 4 were combined due to insufficient enrollment for genotype 4.
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 24
Description: Safety population includes all enrolled participants
Arm/Group | Pegylated Interferon Alfa 2a (Peginterferon)
Serious Adverse Events (participants affected / at risk) | 50/1013
Other Adverse Events (participants affected / at risk) | 131/1013
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon Alfa 2a (Peginterferon) (N=1013)
Anemia (Blood and lymphatic system disorders) | 8
Haemolytic anemia (Blood and lymphatic system disorders) | 1
Neutropenic fever (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Optic nerve disorder (Eye disorders) | 1
Optic Neuropathy (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Asthenia (General disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Abdominal wall abcess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Infection (Infections and infestations) | 1
Tubo-ovarian abcess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Foot fracture (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral hemorrhage (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Major depression (Psychiatric disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Scrotal swelling (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Anal spincterotomy (Surgical and medical procedures) | 1
Hernia repair (Surgical and medical procedures) | 1
Inguinal hernia repair (Surgical and medical procedures) | 1
Sigmoidectomy (Surgical and medical procedures) | 1
Post thrombotic syndrome (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon Alfa 2a (Peginterferon) (N=1013)
Anemia (Blood and lymphatic system disorders) | 103
Neutropenia (Blood and lymphatic system disorders) | 57
Asthenia (General disorders) | 103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.